CLINICAL TRIAL: NCT00840528
Title: Genetic Susceptibility TO Ozone-induced Bronchial Airway Inflammatory Responses In Humans
Brief Title: Genetic Susceptibility TO Ozone-induced Airway Inflammation in Humans
Acronym: GARBOZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 02-1416; NIH/NIEHS 1RC1ES018417 (Other Grant/Funding Number: NIEHS & EPA)
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Healthy Control
Keywords: ozone
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ozone exposure (Experimental): Exposure to ozone at 0.4ppm
  Interventions: Other: ozone

INTERVENTIONS:
Other: ozone — 0.4 ppm ozone for 2 hours
  Other Names: O3

SUMMARY:
The principal purpose of this study is to identify hyper-responsive, responsive and non-responsive groups of healthy human subjects based on their airway neutrophilic response to ozone exposure, and to perform micro-array analyses on DNA collected from recovered airway cells to explore possible differences in gene expression profiles between the three groups

DETAILED DESCRIPTION:
Sputum assessment day: Subjects meeting the required health status following the medical screening will be provided with a verbal and written description of all experimental procedures and possible risks involved in their participation. All subjects will be required to provide written informed consent to participate in the study. The ability of subjects to produce adequate induced sputum samples will also be determined. Therefore the subjects will be asked to produce sputum following inhalation of hypertonic saline (3, 4 and 5%). Subjects should be able to produce at least 50 mg of sputum (selected plug) per sample. Each sputum sample must contain a total cell count of at least 100,000 cells, a differential cell count containing less than 40% squamous epithelial cells, and cell viability of at least 50%, thus minimizing variability in cell recovery and squamous cell contamination. Subjects who are effective sputum producers will then be scheduled for a training session. Subjects may still be excluded from the study if unable to perform adequate pulmonary function tests.

Training session: Training session will occur no less than 2 days prior to exposure

* Lung function tests, including spirometry and plethysmography (body box measurements).
* Introduction to the ozone exposure chamber.
* Instruction on how to use the treadmill, including a minute ventilation measurement to reach the level of exercise required for the study.
* Nitric oxide measurement - this measures the amount of nitric oxide (NO) present in expired air. An increased concentration of NO in exhaled air may be found in normal persons with acute inflammation during upper respiratory tract infections and in association with symptoms in patients with allergic rhinitis. Thus, measurement of the concentration of NO in expired air may be useful as an indirect assessment of airway inflammation. Lung production of NO will be measured by collection of a sample of exhaled gas. Nasal production of NO will be measured directly by connecting a NO analyzer sampling line to one nostril with the other nostril open to ambient air. During the nasal measurement the subject will exhale through a cardboard, disposable tube with a resistance in order to close the palate and prevent contamination of the nasal sample with. The entire procedure should be completed in less than 15 minutes.

Exposure and testing protocol: Upon arrival at the laboratory, subjects' clinical health status will be ascertained by medical personnel, including base line heart rate, blood pressure, evaluation of respiratory symptoms (breath sounds) and general health. All female subjects will be required to provide a menstrual cycle history and a urine sample will be required for pregnancy testing. Each pregnancy test will be considered valid for 7 days. Testing will be postponed if a subject exceeds previously established limits.

The 0.4 ppm ozone exposure will be conducted in an ozone exposure chamber. Each subject will be exposed to ozone for 2 hours. During the exposure, subjects will perform four 15 minute bouts of moderate exercise (minute ventilation or VE = 30 40 L/min) on a treadmill, each separated by 15 minutes of seated rest. Before and after exposure, lung function and breath sounds will be assessed for any signs of bronchial constriction. Venipuncture (as noted above) will occur prior to exposure. Measurements of cardiorespiratory performance will be obtained during each exercise period.

Approximately 4-6 hours following ozone exposure, venipuncture will occur. Subjects will perform the sputum induction procedures described above with nebulized inhaled hypertonic saline (3, 4 and 5%). The subject will remain under medical supervision until pulmonary function (spirometry) returns to within 5% of pre-exposure baseline values before leaving the laboratory. Approximately 24 hours after the ozone exposure, subjects will return to the laboratory for lung function testing and sputum induction, in addition to a venous blood sample.

At each time point (pre and post exposure, and 24 hours post exposure), blood will be drawn from the vein in forearm into clinical lab tubes. During one of these blood draws the additional 5ml will be drawn for genotyping. Plasma will be separated from 4 ml and frozen at 70 degrees C for future analysis of mediators of interest, such as cytokines, as well as other systemic effects of ozone. The remaining blood will be assessed by whole blood assays for markers of inflammatory and immune activation (CD11b, CD14, CD64, CD16, HLA-DR, CD45, CD3, CD80, CD86) and function (phagocytosis and oxidative burst) by two colour flow cytometry. RNA will be extracted from sputum inflammatory cells for microarray analysis,.

During the course of participation all subjects will be required to abstain from; ingestion of Vitamins C and E, aspirin or any other anti-inflammatory medication, exposure to cigarette smoke or other irritants. In addition, subjects will be asked to have nothing by mouth for 2 hours before sputum induction. They will be asked to arrive in the research lab NPO x 2 hours on training day and post exposure day, and will have lunch on exposure day at a time that will allow for the 2 hour NPO requirement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will have an FEV1/FVC equal to or greater than 75%, as well as FVC and FEV1 greater than or equal to 80% of predicted normal for height and age.
* Skin testing will be performed; subjects with active allergies will not be studied while they are symptomatic.
* Subjects must be in good general health with no history of acute or chronic cardiovascular disease, chronic respiratory disease, and acute respiratory illness within 4 weeks, and without contraindications for performing sustained light to moderate exercise.
* Subjects must demonstrate the ability to produce an acceptable induced sputum sample during the training session. If the sample is unsatisfactory, the subject's participation will end at this point.
* Antidepressants and other medications may be permitted if in the opinion of the investigator the medication will not interfere with the study procedures or compromise safety; and if the dosage has been stable for 3 months.
* Subjects must smoke less than 10 cigarettes (one half pack) a month for at least 3 years. Individuals who have smoked greater than 10 pack years lifetime will be excluded.
* Subjects must be willing to refrain from strenuous physical activity for 24 hours before and after exposure.

Exclusion Criteria:

* asthmatic or active allergic rhinitis
* Non English speaking volunteers will be excluded as no one on the study staff is fluent in other languages likely to be encountered.
* use anti-inflammatory medications or medications for asthma

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2002-02; Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Airway neutrophilic response to ozone exposure | 6-24 hours post challenge

SECONDARY OUTCOMES:
expression of specific genes of interest in a subset of ozone-responsive and ozone-non-responsive subjects | pre/ post exposure

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, MS, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- US EPA Human Studies Facility, Chapel Hill, North Carolina, United States